CLINICAL TRIAL: NCT04995679
Title: Residual Pain After Successful Implant of Metaphyseal Sleeves in Total Knee Arthroplasty: a Case Series of 50 Patients With Long-term Follow-up
Brief Title: Residual Pain After Successful Implant of Metaphyseal Sleeves in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pietro Randelli, MD, Professor, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sleeve
Record Dates: First submitted 2021-05-20; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient whit osteoarthritis of the knee (Other): Patients with osteoarthritis of the knee undergoing total knee replacement surgery with metaphyseal sleeves
  Interventions: Procedure: Implant of metaphyseal sleeves in Total knee arthroplasty

INTERVENTIONS:
Procedure: Implant of metaphyseal sleeves in Total knee arthroplasty — Implant of metaphyseal sleeves in Primary and revision TKA

SUMMARY:
: Total knee revision arthroplasty is increasing in daily practice and will become more relevant in the years to come. Bone loss is a significant challenge in total knee arthroplasty (TKA) especially in revision procedures. Metaphyseal sleeves are widely used to bypass bone loss and improve stability. This study aims to report the results of primary and revision TKA (R-TKA) using metaphyseal sleeves.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they were older than 18 years and underwent a primary or revision TKA using cement-less metaphyseal sleeves, performed by the same senior surgeon

Exclusion Criteria:

* Patients were excluded from the final analysis if they did not have 18 months of minimum follow-up and if they were lost to the final control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of implant's survivorship | 7 years
  A retrospective study was performed on patients who underwent TKA or Revision TKA using tibial and/or femoral metaphyseal sleeves to evaluate the implant's survivorship

SECONDARY OUTCOMES:
Evaluation of Numerical Rating Scale (NRS) | 7 years
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. 0-10 where 0 is no pain and 10 is the worst pain imaginable
Evaluation of Western Ontario and Mc Master University (WOMAC) | 7 years
  The WOMAC is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  A sum of the scores for all three subscales gives a total WOMAC score
Evaluation of Oxford Knee Score (OKS) | 7 years
  The Oxford Knee Score (OKS) is a 12-item patient-reported PRO specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty). It is short, reproducible, valid and sensitive to clinically important changes.
  Each of the 12 answers are assigned the previously defined number of points. They range from 1 = least difficult to 5 = most difficult. The 12 ratings are then added together to give a total score used to assess the patient. The possible total score ranges from 12 to 60 points. Here, a low score (e.g. 12 points) indicates good outcomes and vice versa.

CONTACTS AND LOCATIONS:
Locations (1):
- 2) 1° Clinica Ortopedica, ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO, Milan, Milan, Italy